CLINICAL TRIAL: NCT04863404
Title: Evaluation of the Treatment Effects of Tooth Borne Versus Bone-anchored Protraction Procedures in Class III Patients With Maxillary Deficiency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Burçin Akan, Assistant Professor, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-TDU-DİŞF-0003
Record Dates: First submitted 2021-04-21; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Anterior Crossbite; Class III Malocclusion; Maxillary Deficiency
Keywords: maxillary protraction; tooth-borne vs bone-anchored; face mask; AltRamec; rme; Temporary anchorage devices (TADs) in the anterior palate; hybrid hyrax
MeSH Terms: conditions — Malocclusion, Angle Class III; Retrognathia; Tietz syndrome | interventions — Masks

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: 3 arm parallel clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bone-anchored maxillary protraction group (Experimental): Face mask with hybrid-hyrax
  Interventions: Other: Face mask with hybrid-hyrax
- Tooth-borne maxillary protraction group (Experimental): Face mask with conventional bonded RME
  Interventions: Other: Face mask with conventional bonded RME
- Control group (No Intervention): Control group consisting of 14 non-treated Class III malocclusion subjects

INTERVENTIONS:
Other: Face mask with hybrid-hyrax — Face mask with hybrid-hyrax
  Arms: Bone-anchored maxillary protraction group
Other: Face mask with conventional bonded RME — Face mask with conventional bonded RME
  Arms: Tooth-borne maxillary protraction group

SUMMARY:
The aim of this prospective randomized controlled clinical study is to compare the effects of bone-anchored and tooth borne maxillary protraction on dentofacial structures in skeletal Class III patients.

DETAILED DESCRIPTION:
Today, the treatment of class III malocclusion is becoming more important due to the increased awareness of people about their appearance and the impact of appearance on the psychosocial state.

Various studies have shown that 40% of class III malocclusions are clinically caused by maxillary deficiency, 42% by mandibular excess, and 18% by a combination of maxillary deficiency and mandibular excess.

The face mask is the most effective treatment modality for class III malocclusions caused by a maxillary deficiency. The rationale for using a face mask is to apply heavy forces to the midface to advance the maxilla forward. These forces cause disarticulation by initiating resorption and apposition in the sutural articulations. However, undesirable dental effects arise from the use of tooth-borne rapid maxillary expansion (RME) during these treatments. These include loss of anchorage and incisor proclination during the mesialization of the maxillary dentition, extrusion of the upper molars and posterior mandibular rotation, and insufficient anterior displacement of the maxilla (1-3 mm).

Studies have shown that increasing the skeletal effects can reduce post-treatment relapse, one of the most important problems in orthodontics.

To increase the amount of maxillary skeletal advancement and to minimize the side effects of tooth-borne maxillary expansion and protraction, a new bone-anchored hybrid hyrax appliance has been proposed. Hybrid hyrax treatment has the following advantages over tooth-borne mechanics:

* Since the force is applied close to the center of resistance of the maxilla, counterclockwise rotation of the maxilla and related posterior mandibular rotation are not observed.
* Transversal forces are applied to premolars or deciduous molars and mini implants without the risk of periodontal damage, fenestration, and dehiscence that may occur with tooth-borne appliances are avoided.
* Mesial migration of the dentition, proclination of the upper incisors, and occupation of the necessary place for the canines to erupt are avoided.
* Treatment is minimally invasive.
* Upper and lower arches remain completely accessible for orthodontic interventions.
* Only skeletal maxillary advancement is achieved. In our study, additionally, the Alternate Rapid Maxillary Expansion and Constriction (AltRamec) protocol, which increases the skeletal effects during maxillary protraction by providing more effective disarticulation of circummaxillary sutures than conventional rapid maxillary expansion was used.

ELIGIBILITY:
Inclusion Criteria:

* Late mixed or early permanent dentition
* C3 or C4 period according to the cervical vertebral maturation method
* Presence of skeletal class III malocclusion (ANB <0 °).
* Retrusive nasomaxillary complex (Nperp-A <1 mm).
* Presence of dental class III malocclusion
* Normal or horizontal growth pattern (SNGoGn <40 °).
* Negative overjet (overjet <0)
* Good cooperation
* Absence of any systemic disease
* Periodontal health
* No previous orthodontic treatment
* No craniofacial deformity
* No neuromuscular deformity
* The absence of a congenital anomaly

Exclusion Criteria:

* Poor cooperation
* Early mixed dentition
* Individuals who have passed the C4 period
* Craniofacial deformity
* Congenital anomaly
* A history of facial trauma Syndromes such as cleft lip and palate

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-05-20 (Estimated); Study Completion 2021-10-20 (Estimated)

PRIMARY OUTCOMES:
Pre-treatment (T0) cephalometric analysis measures | 0 month
  A cephalometric analysis of skeletal maxillary (SNA) and mandibular (SNB) positions
Pre-treatment (T0) soft tissues measurements | 0 month
  Maxillary and mandibular (Soft tissue convexity angle) soft tissue analysis using 3D stereophotogrammetry

SECONDARY OUTCOMES:
Post-treatment (T1) cephalometric analysis measurements | An average of 6 month
  Evaluation of pos-treatment cephalometric changes of skeletal maxillary (SNA) and mandibular (SNB) positions
Post-treatment (T1) soft tissues measurements | An average of 6 month
  Evaluation of maxillary and mandibular soft tissue changes (Soft tissue convexity angle) using 3D stereophotogrammetry

CONTACTS AND LOCATIONS:
Overall Officials: Burcin AKAN, Phd, Study Director — Academician
Locations (1):
- Izmir Katip Celebi University,Faculty of Dentistry, Department of Orthodontics, Izmir, Çiğli, Turkey (Türkiye)